CLINICAL TRIAL: NCT00041041
Title: A Phase II Evaluation Of Gleevec (Imatinib Mesylate) (IND #61135, NSC #716051) In The Treatment Of Persistent Or Recurrent Epithelial Ovarian Or Primary Peritoneal Carcinoma
Brief Title: Imatinib Mesylate in Treating Patients With Persistent or Recurrent Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02473; GOG-0170E; U10CA027469 (NIH); CDR0000069438 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have persistent or recurrent ovarian epithelial or primary peritoneal cancer. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the cytostatic, anti-tumor activity of Gleevec (Imatinib Mesylate) through the probability of surviving progression-free for at least 6 months in patients with recurrent or persistent epithelial ovarian or primary peritoneal carcinoma receiving Gleevec.

II. To determine the frequency and severity of adverse effects of Gleevec in this cohort of patients as assessed by CTC.

SECONDARY OBJECTIVES:

I. To determine the distribution of the overall survival. II. To determine the distribution of progression-free survival. III. To estimate the clinical response rate (partial and complete response as defined under the RECIST criteria).

IV. To assess the effects of prognostic variables: initial performance status, platinum sensitivity, and mucinous (or clear cell) histology).

TERTIARY OBJECTIVES:

I. To determine the levels of expression of c-KIT and its ligand, stem cell factor (SCF) in archived, formalin fixed, paraffin embedded primary tumors collected prior to the initiation of first-line chemotherapy.

II. To determine the levels of expression of platelet derived growth factor receptor (PDGFR) and its ligand PDGF in archived, formalin fixed, paraffin embedded primary tumors collected prior to the initiation of first-line chemotherapy.

III. To determine the levels of expression of AKT2 and its activated form, phospho-AKT2, in archived, formalin fixed, paraffin embedded primary tumors collected prior to the initiation of first-line chemotherapy.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma

  * Recurrent or persistent disease
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Tumors within a previously irradiated field considered nontarget lesions
* At least one prior platinum-based chemotherapy regimen (containing carboplatin, cisplatin, or another organoplatinum compound) for primary disease required

  * Initial treatment may include high-dose, consolidation, or extended therapy
  * Initial treatment-free interval less than 12 months for patients who received only 1 prior platinum-based regimen
  * Initial treatment-free interval of more than 12 months allowed provided disease progression has occurred within 12 months after retreatment with a second-line platinum-based regimen
* Ineligible for a higher priority GOG protocol (e.g., any active phase III GOG protocol for the same patient population)
* Performance status - GOG 0-2 (if patient has received one prior treatment regimen)
* Performance status - GOG 0-1 (if patient has received two prior treatment regimens)
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No active infection requiring antibiotics
* No greater than grade 1 sensory and motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No signs or symptoms of bowel dysfunction
* At least 3 weeks since prior immunologic therapy directed at the malignant tumor
* No concurrent biologic therapy or immunotherapy for the malignant tumor
* Recovered from prior chemotherapy
* No prior noncytotoxic chemotherapy for persistent or recurrent disease
* One additional cytotoxic regimen for persistent or recurrent disease allowed
* No concurrent chemotherapy for the malignant tumor
* At least 1 week since prior hormonal therapy directed at the malignant tumor
* No concurrent therapeutic corticosteroids
* No concurrent anticancer hormonal therapy
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* No prior radiotherapy to more than 25% of marrow-bearing areas
* No concurrent anticancer radiotherapy
* Recovered from recent prior surgery
* At least 3 weeks since other prior therapies directed at the malignant tumor
* No prior imatinib mesylate
* No prior anticancer therapy that would preclude study participation
* No concurrent therapeutic anticoagulation with warfarin
* No other concurrent investigational drugs
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-06; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | At 6 months
Frequency and severity of adverse effects as assessed by CTC | Up to 7 years

SECONDARY OUTCOMES:
Duration of overall survival | Up to 7 years
Duration of progression-free survival | Up to 7 years
Frequency of clinical response (partial and complete response) | Up to 7 years
Prognostic variables: initial performance status, age, platinum sensitivity, and mucinous (or clear cell) histology | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States